CLINICAL TRIAL: NCT04584463
Title: Factors Associated With Neurological Prognosis 30 Days After an ICU Admission for a Myocardial Infarction Complicated by an Out-of-Hospital Cardiac Arrest : an Observationnal Multicentric Study
Brief Title: Factors Associated With CPC 1-2 in 110 Patients Admitted in French ICU for a Myocardial Infarction Complicated by an OHCA.
Acronym: ACR-MI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Bruno LEVY, Professor Bruno LEVY, Central Hospital, Nancy, France
Other Study IDs: 2019PI166
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Myocardial Infarction; Coma; Outcome, Fatal; Neurologic Dysfunction
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Myocardial Infarction; Coma; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluate the association of some in-ICU factors with the neurological prognosis of patients admitted for an out-of-hospital cardiac arrest due to a myocardial infarction.

DETAILED DESCRIPTION:
Pre-hospital factors associated with poor neurologic outcome are well known. Meanwhile, in-ICU factors for the first 24 hours may impact neurologic outcome.

This observational study aim to study the factors such as ECLS, NSE dosage, therapeutic hypotermia... and their association with neurologic outcome in patient with myocardial infarction due to instable coronaropathy complicated by an out-of-+hospital cardiac arrest.

This is designed to be a observationnal, prospective, multicentric national french study

ELIGIBILITY:
Inclusion Criteria:

* aged of 18 years old or more
* non opposition of the patient, or his family if he is unable to consent, after loyal and comprehensive explanation
* patient admitted in ICU
* the reason for admission is a resurected out-of-hospital cardiac arrest
* the cause of the cardiac arrest is a type 1 myocardial infarction

Exclusion Criteria:

* refractory cardiac arrest (no flow > 30 minutes in normothermia)
* in-hospital cardiac arrest
* pregnancy
* patient under juridic protection
* opposition of the patient, or of his family is he is unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient older than 18 years old admitted in an ICU following resurected out-of-hospital cardiac arrest due to a type 1 myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Neurologic outcome (CPC) | 30 day from in-ICU admission
  Cerebral Performance Category Scale to assess neurologic outcome 1-2 : good outcome 3-4-5 : bad outcome

SECONDARY OUTCOMES:
Neurologic outcome (Rankin) | 30 day from in-ICU admission
  Rankin score to assess neurologic outcome
  * 0-1-2 good outcome
  * 3-4-5 bad outcome
death | 30 day form in-ICU admission
  all-causes death

IPD SHARING:
Plan to Share IPD: No